CLINICAL TRIAL: NCT06447129
Title: Effect of NMES as an Add-On to Exercise Program in Degenerative Meniscus Tears: A Randomized Controlled Trial
Brief Title: Effect of NMES as an Add-On to Exercise Program in Degenerative Meniscus Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 216
Record Dates: First submitted 2024-06-03; First posted 2024-06-06 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-06

CONDITIONS: Degenerative Disease; Meniscus Tear; Knee Pain Swelling
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMES with Exercise (Experimental): Each subject in Group 2 will receive a treatment protocol consisting of stretching exercises, strengthening exercises, functional exercises for the knee and hip, and NMES application for the quadriceps femoris muscle.
  Interventions: Other: Exercise; Other: Neuromuscular electrical stimulation
- Exercise (Active Comparator): Each subject in Group 2 will receive a treatment protocol consisting of stretching exercises, strengthening exercises, functional exercises for the knee and hip.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — An 8-week exercise program used in conservative treatment of degenerative meniscus tears will be performed.
  The patients will do exercises under the control of the physiotherapist in the clinic.
  The patient will perform the exercises with the verbal and visual commands of the physiotherapist.
Other: Neuromuscular electrical stimulation — The Neuromuscular Electrical Stimulation (NMES) will be applied for 20 minutes. The patient will be seated with hips and knees flexed at 90°. Electrodes will be placed on the proximal and distal ends of the vastus medialis obliquus and vastus lateralis muscles. The intensity will be increased as much as the patient can tolerate, and the patient will be asked to relax and not make voluntary muscle contractions.
  Arms: NMES with Exercise

SUMMARY:
This randomized-controlled trial aims to investigate the effect of NMES as an add-on to an exercise program in patients with degenerative meniscus tears.

DETAILED DESCRIPTION:
To investigate the efficacy of NMES as an add-on to an exercise program, voluntary patients with degenerative meniscus tears, aged between 40 and 65 years, will be randomly divided into two groups: Group 1 (NMES with Exercise) and Group 2 (Exercise). Interventions will be applied for 16 sessions (twice a week for 8 weeks). The patients will be assessed at baseline and at the end of the 8-week intervention. The pain during activity, at rest, and at night will be assessed with the Visual Analog Scale (VAS). Active range of motion will be assessed with a digital goniometer. Isometric muscle strength will be measured with a handheld dynamometer. The functional status and symptoms will be evaluated by the Knee Injury and Osteoarthritis Outcome Score (KOOS) and Lysholm Knee Scoring Scale. Health-related quality of life will be assessed with the Short Form-12 (SF-12).

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 40 and 65 years
* Having the degenerative meniscus tear in at least one knee
* Having body mass index in the range of 18-30 kg/m2
* Feeling the pain that lasts for at least 2 months
* Having grade 1 or grade 2 degenerative meniscal tear diagnosed by an orthopedic specialist according to the MRI results
* Having the ability to read and write Turkish

Exclusion Criteria:

* Having undergone arthroscopic partial meniscectomy surgery due to degenerative meniscal tear
* Participating in a physiotherapy program for degenerative meniscal tear in the last 12 weeks
* Have received steroid injections in the last 6 months
* Accompanying conditions such as injury to the surrounding ligaments, congenital anomaly in the affected knee, coxarthrosis and spinal stenosis
* Presence of any systemic disorder that may affect assessment parameters
* Failure to cooperate with assessments

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline
  Short-term and long-term symptoms and function will be assessed with the Knee injury and Osteoarthritis Outcome Score (KOOS) that is developed as an extension of the WOMAC Osteoarthritis Index. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At the end of 8-week intervention
  Short-term and long-term symptoms and function will be assessed with the Knee injury and Osteoarthritis Outcome Score (KOOS) that is developed as an extension of the WOMAC Osteoarthritis Index. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Visual Analogue Scale (VAS) | Baseline
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Visual Analogue Scale (VAS) | At the end of 8-week intervention
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Active Range of Motion | Baseline
  Active knee range of motion including flexion and extension will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a digital goniometer.
Active Range of Motion | At the end of 8-week intervention
  Active knee range of motion including flexion and extension will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a digital goniometer.
Muscle Strength | Baseline
  Isometric muscle strength will be measured with a handheld dynamometer for knee flexors and extensors. The process will be repeated three times in each direction, with the average value recorded.
Muscle Strength | At the end of the 8-week intervention
  Isometric muscle strength will be measured with a handheld dynamometer for knee flexors and extensors. The process will be repeated three times in each direction, with the average value recorded.
Lysholm Score | Baseline
  Functional limitations related to degenerative meniscal tear will be used with the Lysholm Score that is one of the most frequently used functional questionnaires. The total score is the sum of each response to the eight questions, and may range from 0-100. Higher scores indicate a better outcome with fewer symptoms or disability.
Lysholm Score | At the end of the 8-week intervention
  Functional limitations related to degenerative meniscal tear will be used with the Lysholm Score that is one of the most frequently used functional questionnaires. The total score is the sum of each response to the eight questions, and may range from 0-100. Higher scores indicate a better outcome with fewer symptoms or disability.
Short Form-12 (SF-12) | Baseline
  Short Form-12 (SF-12), which is developed based on Short Form-36, consists of 12 items: 7 items dealing with the physical components scores (PCS-12) and 5 items related to the mental components scores (MCS-12) of SF-12. Range of both scores is 0 to 100, where the higher scores indicate better health related quality of life.
Short Form-12 (SF-12) | At the end of the 8-week intervention
  Short Form-12 (SF-12), which is developed based on Short Form-36, consists of 12 items: 7 items dealing with the physical components scores (PCS-12) and 5 items related to the mental components scores (MCS-12) of SF-12. Range of both scores is 0 to 100, where the higher scores indicate better health related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)